CLINICAL TRIAL: NCT03126435
Title: A Randomized Controlled, Open Label, Adaptive Phase-3 Trial to Evaluate Safety and Efficacy of EndoTAG-1+GEM vs GEM Alone in Patients With Measurable Locally Advanced/Metastatic Adenocarcinoma of the Pancreas Failed on FOLFIRINOX Treatment
Brief Title: EndoTAG-1+GEM vs GEM in Patients With Locally Advanced/Metastatic Pancreatic Adenocarcinoma Failed on FOLFIRINOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SynCore Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT4006
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Pancreas Cancer; Locally Advanced Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: FOLFIRINOX; 5-Fluorouracil; folinic acid; irinotecan; oxaliplatin; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — MBT-0206; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EndoTAG-1 and Gemcitabine (Experimental): EndoTAG-1 22 mg/m² twice weekly plus Gemcitabine 1000mg/m² once weekly for 1 cycle (8 weeks) consisting of 3 weeks of treatment and 1 week rest followed by 3 weeks of treatment and 1 week rest until any one of the following occurs: progressive disease or unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: EndoTAG-1; Drug: Gemcitabine
- Gemcitabine Monotherapy (Active Comparator): Gemcitabine 1000mg/m² once weekly, for 1 cycle (8 weeks) consisting of 3 weeks of treatment and 1 week rest followed by 3 weeks of treatment and 1 week rest until any one of the following occurs: progressive disease or unacceptable toxicity or withdrawal of consent.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: EndoTAG-1 — twice weekly
  Other Names: EndoTAG-1 was first developed by Munich Biotech AG (Germany) under the names LipoPac and MBT-0206 and by Medigene AG under the name of EndoTAG-1.
  Arms: EndoTAG-1 and Gemcitabine
Drug: Gemcitabine — once weekly
  Other Names: Gemcitabine Hydrochloride

SUMMARY:
The aim of this adaptive Phase 3 trial is to show a statistically significant superiority of EndoTAG-1 in combination with gemcitabine compared to gemcitabine monotherapy in patients with locally advanced/metastatic pancreatic cancer after FOLFIRINOX failure.

DETAILED DESCRIPTION:
The objective of the study was to assess the safety and efficacy of a combination therapy of EndoTAG-1 plus gemcitabine vs. gemcitabine monotherapy in patients with locally advanced and/or metastatic adenocarcinoma of the pancreas eligible for second-line therapy after failing first line therapy with FOLFIRINOX

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Written informed consent
3. Histologically or cytologically confirmed adenocarcinoma of the pancreas
4. Metastatic or locally advanced disease that is considered unresectable
5. Measurable / assessable disease according to RECIST v.1.1
6. Documented disease progression on first line FOLFIRINOX
7. Negative pregnancy test
8. Both male and female patients and their partners of childbearing potential must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, tubal sterilization or vasectomy) or must practice complete abstinence from intercourse of reproductive potential during the course of the study and for 90 days after last treatment (excluding women who are not of childbearing potential and men who have been sterilized).
9. ECOG performance status 0 or 1

Exclusion Criteria:

1. Cardiovascular disease, New York Heart Association (NYHA) III or IV
2. History of severe supraventricular or ventricular arrhythmia
3. History of coagulation or bleeding disorder
4. History of acute myocardial infarction within 6 months before randomization
5. History of congestive heart failure
6. Acute or chronic inflammation (autoimmune or infectious)
7. Significant active/unstable non-malignant disease likely to interfere with study assessments
8. Laboratory tests (hematology, chemistry) outside specified limits:

   1. WBC ≤ 3 x 10³/mm³
   2. ANC ≤ 1.5 x 10³/mm³
   3. Platelets ≤ 100.000/mm³
   4. Hb ≤ 9.0 g/dl (≤ 5.6 mmol/l)
   5. aPTT > 1.5 x ULN
   6. Serum creatinine > 2.0 mg/dl (> 176.8 μmol/l)
   7. AST and/or ALT > 2.5 x ULN; for patients with significant liver metastasis AST and/or ALT > 5 x ULN
   8. Alkaline phosphatase > 2.5 x ULN
   9. Total bilirubin > 2 x ULN
   10. Albumin < 2.5 g/dL
9. Clinically significant ascites
10. Any anti-tumor treatment (except FOLFIRINOX as the first-line therapy) for pancreatic adenocarcinoma before enrollment. Note: Patients who have undergone surgical interventions for pancreatic adenocarcinoma will be eligible.
11. Any radiotherapy for pancreatic adenocarcinoma before enrollment except for treatment of bone metastases if target lesions are not included in the irradiated field
12. Major surgery < 4 weeks prior to enrollment
13. Pregnant or nursing
14. Investigational medicinal product < 4 weeks of enrollment
15. Documented HIV history
16. Active hepatitis B infection requiring acute therapy Note: Subjects infected by the hepatitis B virus will be eligible for the study if they have no signs of hepatic decompensation and meet the liver function tests eligibility criteria.
17. Known hypersensitivity to any component of the EndoTAG-1 and/or gemcitabine formulations
18. History of malignancy other than pancreatic cancer < 3 years prior to enrollment, except nonmelanoma skin cancer or carcinoma in situ of the cervix treated locally
19. Vulnerable populations (e.g. subjects unable to understand and give voluntary informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Ph.D., Principal Investigator — National Cheng Kung University Hospital,Tainan, Taiwan, R.O.C
Locations (68):
- United States (16):
  - Compassionate Cancer Care Medical Group, Inc, Corona, California
  - Emory University Hospital, Atlanta, Georgia
  - John B. Amos Cancer Center / IACT Health, Columbus, Georgia
  - Orchard Healthcare Research (OHR) Inc., Skokie, Illinois
  - Investigator Clinical Research Centers of Indiana, Indianapolis, Indiana
  - Cotton O'Neil Cancer Center (Stormont-Vail Cancer Center), Topeka, Kansas
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - North Mississippi Hematology & Oncology Associates, Ltd., Tupelo, Mississippi
  - Southeast Nebraska Cancer Center (SNCC) - Central Clinic - Main Clinic, Lincoln, Nebraska
  - Guthrie - Corning Hospital - Guthrie Cancer Center, Sayre, Pennsylvania
  - Charleston Cancer Center, North Charleston, South Carolina
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Scott & White Vasicek Cancer Treatment Center, Temple, Texas
  - Renovatioclinical, The Woodlands, Texas
  - University of Virginia Hospital, Charlottesville, Virginia
- France (15):
  - CHU Angers, Angers
  - CHRU - Besançon, Besançon
  - Hopital Haut Leveque, Bordeaux
  - CHRU Brest - Hôpital Morvan, Brest
  - Centre Hospitalier de Cholet, Cholet
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - Hôpital Privé Jean Mermoz, Lyon
  - La Timone, Marseille
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Antoine-Lacassagne, Nice
  - Hopital La Pitié Salpétrière, Paris
  - CH Saint Jean, Perpignan
  - Centre Eugène Marquis, Rennes
  - Clinique Sainte Anne/Strasbourg Oncologie Leberale, Strasbourg
- Hungary (6):
  - Dél-pesti Centrumkórház - Országos Hematológia és Infektológia Intézet, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Bács-Kiskun Megyei Kórház Onkoradiológiai Központ, Kecskemét
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Pécsi Tudomány Egyetem Onkoterápiás Intézet, Pécs
- Israel (5):
  - Oncology Department, Hillel Yafe MC, Hadera
  - Rambam Health Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Russia (7):
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - Kursk State Clinical Oncology Dispensary, Kursk
  - Federal State Budgetary Scientific Institution "Russian Oncological Scientific Center named after N.N.Blokhin", Moscow
  - Private clinnic "Medicine 24/7", Moscow
  - Budget Institution of Healthcare of Omsk Region "Clinical Oncology Dispensary", Omsk
  - State Budget Healthcare Institution "Orenburg Region Clinical Oncological Dispensary", Orenburg
  - State Budgetary Healthcare Institution Leningrad Regional Oncology Center, Saint Petersburg
- South Korea (9):
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Inha University Hospital, Incheon
  - Chonnam National University Hwasun Hospital, Jeongnam
  - CHA Bundang Medical Center, Seongnam
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Medical Foundation - Kaohsiung Branch, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital-Taipei Branch, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital (TSGH), Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 218 subjects were enrolled between October 2018 and July 2020.
Groups:
- EndoTAG-1 and Gemcitabine: EndoTAG-1 22 mg/m² twice weekly plus Gemcitabine 1000 mg/m² once weekly for 1 cycle (8 weeks) consisting of 3 weeks of treatment and 1 week rest followed by 3 weeks of treatment and 1 week rest until any one of the following occurs: progressive disease or unacceptable toxicity or withdrawal of consent.
  EndoTAG-1: twice weekly
  Gemcitabine: once weekly
- Gemcitabine Monotherapy: Gemcitabine 1000 mg/m² once weekly, for 1 cycle (8 weeks) consisting of 3 weeks of treatment and 1 week rest followed by 3 weeks of treatment and 1 week rest until any one of the following occurs: progressive disease or unacceptable toxicity or withdrawal of consent.
  Gemcitabine: once weekly
Period: Overall Study
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Started | 108 | 110
Completed | 2 | 6
Not Completed | 106 | 104
Not completed — Death | 90 | 84
Not completed — Lost to Follow-up | 4 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 6 | 12
Not completed — e.g. Sponsor Decision, General Deterioration... | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy | Total
Number analyzed (Participants) | 108 | 110 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 72 | 141
  >=65 years | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.98) | 61.7 (9.68) | 61.2 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 50 | 88
  Male | 70 | 60 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 31 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 56 | 59 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  South Korea | 13 | 18 | 31
  Hungary | 15 | 17 | 32
  United States | 6 | 8 | 14
  Taiwan | 21 | 13 | 34
  Israel | 7 | 6 | 13
  France | 20 | 21 | 41
  Russia | 26 | 27 | 53
Extent of Disease at Randomization [Count of Participants; unit: Participants]
  Metastatic | 94 | 95 | 189
  Locally Advanced | 14 | 15 | 29
ECOG Performance at Randomization [Count of Participants; unit: Participants] — ECOG 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 49 | 48 | 97
    1 | 59 | 62 | 121

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The efficacy of EndoTAG-1 treatment was demonstrated through number of events, meaning subject death, compared to number of subjects censored at the time of analysis.
Time Frame: From randomization to death from any cause or last day known to be alive, up to approximately 33.5 months (assessed continuously during treatment)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 108 | 110
days | 226 [183.0 to 278.0] | 209 [158.0 to 248.0]
Statistical Analysis 1: Comparison: EndoTAG-1 and Gemcitabine vs Gemcitabine Monotherapy; Test type: Superiority; p = 0.6647, Log Rank; P-Value is from a stratified log-rank test

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The efficacy of EndoTAG-1 treatment was demonstrated through number of events, meaning first observation of progressive disease, compared to number of subjects censored at the time of analysis.
Time Frame: From randomization to either first observation of progressive disease or occurrence of death, up to approximately 33.5 months (assessed continuously during treatment)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 108 | 110
days | 113 [79.0 to 168.0] | 110 [60.0 to 115.0]
Statistical Analysis 1: Comparison: EndoTAG-1 and Gemcitabine vs Gemcitabine Monotherapy; Test type: Superiority; p = 0.4345, Log Rank; P-Value is from a stratified log-rank test

3. Secondary Outcome: Percentage of Subjects With Objective Response
Description: Percentage of subjects with objective response is based on assessment of complete response (CR) or partial response (PR) according to RECIST v.1.1.
Time Frame: Up to approximately 33.5 months (assessed continuously during treatment)
Population: Of the 108 subjects that received EndoTAG-1 and Gemcitabine, 11 subjects (11.46%, 11/96) presented with a complete or partial response. There were 6 subjects (6.82%, 6/88) that received Gemcitabine Monotherapy considered to have an objective response. For 12 subjects in the EndoTAG-1 group and 22 subjects in the Gemcitabine Monotherapy group, objective response assessments were missing.
Measure: Count of Participants; unit: Participants
Groups:
- EndoTAG-1 and Gemcitabine: EndoTAG-1 22 mg/m² twice weekly plus Gemcitabine 1000 mg/m² once weekly for 1 cycle (8 weeks) consisting of 3 weeks of treatment and 1 week rest followed by 3 weeks of treatment and 1 week rest until any one of the following occurs: progressive disease or unacceptable toxicity or withdrawal of consent.
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 96 | 88
Participants | 11 | 6
Statistical Analysis 1: Comparison: EndoTAG-1 and Gemcitabine vs Gemcitabine Monotherapy; Test type: Superiority; p = 0.2632, Regression, Logistic; P-value is from logistic regression model adjusted for stratification factors among non-missing records

4. Secondary Outcome: Duration of Response
Description: Duration of Response = (date of tumor progression or death - date of first objective response (CR or PR) +1) / 30.
Time Frame: From the first documentation of objective tumor response (date of the first CR or PR) to objective tumor progression or death due to any cause.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 11 | 6
Months | 5.8 (2.62) | 9.1 (6.97)

5. Secondary Outcome: Percentage of Subjects With Disease Control According to RECIST v.1.1
Description: Percentage of subjects with disease control is based on assessment of complete response (CR) or partial response (PR) or stable disease (SD) according to RECIST v.1.1
Time Frame: Up to approximately 33.5 months (assessed continuously during treatment)
Population: There were 12 subjects in the EndoTAG-1 treated group and 22 subjects in the Gemcitabine Monotherapy group that were not included in analysis due to missing records.
Measure: Count of Participants; unit: Participants
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 96 | 88
Participants | 57 | 43
Statistical Analysis 1: Comparison: EndoTAG-1 and Gemcitabine vs Gemcitabine Monotherapy; Test type: Superiority; p = 0.1002, Regression, Logistic; P-value is from logistic regression model adjusted for stratification factors among non-missing records

6. Secondary Outcome: Serum Carcinoma Antigen 19-9 (CA 19-9) Response Rate
Description: Responders are defined as subjects with a reduction in CA 19-9 levels by least 50% from baseline to the end of cycle 1 (or end of full treatment course). If a subject died while on study, he/she was classified as a failure, regardless of previous assessments.
Time Frame: Up to approximately 33.5 months (assessed at baseline, end of cycle 1 or the full treatment course)
Measure: Count of Participants; unit: Participants
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 108 | 110
Participants | 2 | 2
Statistical Analysis 1: Comparison: EndoTAG-1 and Gemcitabine vs Gemcitabine Monotherapy; Test type: Superiority; p = 0.9882, Regression, Logistic; P-value is from logistic regression model adjusted for stratification factors among non-missing records

7. Other Pre Specified Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Pancreatic 26 (EORTC QLQ- PAN26) Score
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Pancreatic 26 (EORTC QLQ- PAN26) consists of 26 questions (Qs) relating to disease symptoms, treatment (Tx) side effects and emotional issues specific to pancreatic cancer (PC). Questions include on altered bowled habits, pain, dietary changes, disease and Tx-related symptoms and issues related to the emotional and social well-being of participants with PC. All 26 Qs are answered on 4-point Likert scale ranging from '1=not at all' to 4='very much' and subsequently transformed into scales that range from 0-100; higher scores= greater degree of symptoms or treatment side effects and emotional issues.
Time Frame: Up to approximately 33.5 months (assessed at baseline and end of treatment (EOT))
Population: Some missing data (Change from baseline is based on subjects with paired values.)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 108 | 110
score on a scale
  Pancreatic pain: number analyzed (Participants) | 60 | 53
  Pancreatic pain | 1.0 (3.0) | 1.7 (3.2)
  Digestive: number analyzed (Participants) | 60 | 53
  Digestive | 0.6 (2.1) | 0.9 (1.6)
  Altered bowel habit: number analyzed (Participants) | 60 | 53
  Altered bowel habit | 0.5 (1.8) | -0.1 (1.5)
  Hepatic: number analyzed (Participants) | 60 | 53
  Hepatic | 0.0 (0.9) | 0.0 (1.1)
  Body image: number analyzed (Participants) | 58 | 54
  Body image | 0.6 (1.8) | 0.7 (1.9)
  Health care satisfaction: number analyzed (Participants) | 59 | 54
  Health care satisfaction | 0.8 (1.6) | 0.4 (1.6)
  Sexuality: number analyzed (Participants) | 57 | 50
  Sexuality | -0.1 (2.4) | 0.8 (2.5)

8. Other Pre Specified Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Core-30 (EORTC QLQ- C30) Score
Description: Change From Baseline in European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Core-30 (EORTC QLQ- C30): included functional scales (physical, role, cognitive, emotional, and social), global health status (GHS), symptom scales (fatigue, pain, nausea/ vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score = better level of functioning or greater degree of symptoms. Change from baseline = Cycle/day score minus baseline score.
Time Frame: Up to approximately 33.5 months (assessed at baseline and end of treatment (EOT))
Population: Some missing data (Change from baseline is based on subjects with paired values.)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EndoTAG-1 and Gemcitabine: EndoTAG-1 22 mg/m2 twice weekly plus Gemcitabine 1000 mg/m² once weekly for 1 cycle (8 weeks) consisting of 3 weeks of treatment and 1 week rest followed by 3 weeks of treatment and 1 week rest until any one of the following occurs: progressive disease or unacceptable toxicity or withdrawal of consent.
  EndoTAG-1: twice weekly
  Gemcitabine: once weekly
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
Number analyzed (Participants) | 108 | 110
score on a scale
  Global health QoL: number analyzed (Participants) | 60 | 54
  Global health QoL | -1.6 (2.7) | -2.0 (2.7)
  Functional scales: number analyzed (Participants) | 60 | 54
  Functional scales | 5.4 (8.2) | 6.9 (9.0)
  Symptom scales: number analyzed (Participants) | 60 | 54
  Symptom scales | 2.6 (4.4) | 2.6 (4.5)
  Side effect scales: number analyzed (Participants) | 60 | 54
  Side effect scales | 1.3 (2.6) | 1.4 (3.0)
  Physical: number analyzed (Participants) | 60 | 54
  Physical | 2.0 (3.1) | 2.4 (3.4)
  Role: number analyzed (Participants) | 60 | 54
  Role | 1.1 (1.7) | 1.4 (1.9)
  Cognitive: number analyzed (Participants) | 60 | 54
  Cognitive | 0.5 (1.2) | 0.6 (1.5)
  Emotional: number analyzed (Participants) | 60 | 54
  Emotional | 1.2 (2.6) | 1.6 (3.0)
  Social: number analyzed (Participants) | 59 | 54
  Social | 0.6 (1.7) | 0.9 (1.6)
  Fatigue: number analyzed (Participants) | 60 | 54
  Fatigue | 1.5 (2.2) | 1.4 (2.1)
  Pain: number analyzed (Participants) | 60 | 54
  Pain | 0.7 (1.8) | 0.9 (2.0)
  Nausea/vomiting: number analyzed (Participants) | 60 | 54
  Nausea/vomiting | 0.4 (1.5) | 0.2 (1.5)
  Dyspnoea: number analyzed (Participants) | 59 | 54
  Dyspnoea | 0.5 (0.9) | 0.6 (0.9)
  Appetite loss: number analyzed (Participants) | 60 | 53
  Appetite loss | 0.5 (1.1) | 0.3 (0.9)
  Insomnia: number analyzed (Participants) | 60 | 53
  Insomnia | 0.0 (0.9) | 0.2 (1.2)
  Constipation/diarrhea: number analyzed (Participants) | 60 | 54
  Constipation/diarrhea | 0.4 (1.2) | 0.4 (1.2)

ADVERSE EVENTS:
Time Frame: Up to approximately 33.5 months (assessed continuously during treatment)
Description: All-Cause Mortality was assessed in all randomized participants. Serious and Other Adverse Events were assessed in the safety population (i.e., subject receiving the treatment after randomization). There were 102 subjects treated with EndoTAG-1 + gemcitabine and 102 subjects treated with gemcitabine monotherapy.
  Systematic Assessment: regular laboratory testing Non-Systematic Assessment: self-reporting by participants or their family members, occasional assessment/testing
Arm/Group | EndoTAG-1 and Gemcitabine | Gemcitabine Monotherapy
All-Cause Mortality (participants affected / at risk) | 91/108 | 85/110
Serious Adverse Events (participants affected / at risk) | 52/102 | 48/102
Other Adverse Events (participants affected / at risk) | 101/102 | 100/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoTAG-1 and Gemcitabine (N=102) | Gemcitabine Monotherapy (N=102)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1)
Death (General disorders) | 0 (0) | 4 (4)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 3 (3)
Malignant biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 1 (2)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoTAG-1 and Gemcitabine (N=102) | Gemcitabine Monotherapy (N=102)
Platelet Count Decreased (Investigations) | 41 (200) | 42 (193)
Neutrophil Count Decreased (Investigations) | 18 (83) | 21 (83)
White Blood Cell Count Decreased (Investigations) | 18 (58) | 17 (71)
Alanine Aminotransferase Increased (Investigations) | 17 (43) | 17 (31)
Aspartate Aminotransferase Increased (Investigations) | 14 (30) | 17 (29)
Gamma-Glutamyltransferase Increased (Investigations) | 11 (19) | 11 (14)
Blood Alkaline Phosphatase Increased (Investigations) | 15 (32) | 5 (9)
Weight Decreased (Investigations) | 13 (19) | 4 (6)
Lymphocyte Count Decreased (Investigations) | 8 (39) | 7 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 2 (3)
Neuropathy Peripheral (Nervous system disorders) | 7 (7) | 4 (5)
Insomnia (Psychiatric disorders) | 9 (10) | 3 (3)
Fatigue (General disorders) | 19 (35) | 16 (22)
Chills (General disorders) | 18 (24) | 6 (12)
Oedema Peripheral (General disorders) | 18 (24) | 6 (12)
Decreased Appetite (Metabolism and nutrition disorders) | 35 (42) | 22 (28)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (13) | 5 (9)
Constipation (Gastrointestinal disorders) | 20 (22) | 20 (24)
Abdominal Distension (Gastrointestinal disorders) | 8 (9) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03126435/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT03126435/SAP_001.pdf